CLINICAL TRIAL: NCT05812846
Title: Monitoring of the Ischemic Stroke Patient Through the Use of New Serum Biomarkers and MRI Imaging
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: 2250
Record Dates: First submitted 2023-03-08; First posted 2023-04-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-03

CONDITIONS: Stroke
Keywords: stroke; biomarkers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this study will be the evaluation (by ELISA quantification and quantitative RT-PCR) of circulating biomarkers of damage and regeneration in patients affected by ischemic stroke. The biomarker levels will be measured from the acute event (48h) and in subsequent 4 times (7 days, 30 days, 90 days, 180 days) following hospitalization, up to 6 months after the acute event. These data will then be correlated for all five times with the clinical scales normally used for patient evaluation and will also be associated with MRI-DTI measurements performed in the post-acute (30 days) and post-discharge (180 days) phase.

DETAILED DESCRIPTION:
In current clinical practice, outcome's assessment after stroke and patients' monitoring during rehabilitation rely on scores in clinical scales and instrumental evaluations (electrophysiological evaluations and MRI imaging). This approach follows current guidelines but has some limitations:

* subjectivity of the patient's clinical evaluation and instrumental data's interpretation
* poor prognostic value of clinical scales;
* poor prognostic value of instrumental measurements;
* difficulty in standardizing and automating clinical/instrumental assessments;
* difficulty in evaluating medical services on a large scale due to the lack of discrete values of treatment efficacy.

The identification and validation of reliable and accessible biomarkers associated with patients' functional recovery could improve their care but still remains a clinical challenge.

Aim of this study will be to measure the levels of circulating biomarkers of brain damage and regeneration in patients affected by ischemic stroke, and to evaluate their prognostic relevance over a 6-month follow-up. Biomarkers' levels will be measured by ELISA and quantitative RT-PCR from the acute event (within 24h from symptoms onset) and in subsequent 4 time-points (7 days, 30 days, 90 days, 180 days post-stroke). Obtained data will be correlated with clinical scales used for patient evaluation and will be associated with MRI-DTI measurements performed in the post-acute (30 days) and post-discharge (180 days) phase.

ELIGIBILITY:
Inclusion Criteria:

* First occurrence of brain injury, confirmed on CT imaging, determined by ischemic stroke
* Patient able to sign an informed consent, alternatively legal representative or relative

Exclusion Criteria:

* Previous ischemic events
* Previous head trauma of any entity
* New onset of acute events during the study
* Previous illness, diagnosis or suspicion of current illness with central nervous system involvement
* Diagnosis of cognitive impairment prior to the acute event (MMSE < 24)
* Need for walking assistance prior to the acute event
* Diagnosis of autoimmune diseases
* Diagnosis of haematological or oncological disease
* Diagnosis of a psychiatric condition: bipolar disorder, psychosis, schizophrenia or suicidal ideation
* Subjects with relative and absolute contraindications to magnetic resonance imaging.
* Life expectancy less than 1 year
* Dependence or abuse of alcohol, drugs or psychotropics prior to the acute event
* Pregnancy in progress
* Severe renal or hepatic insufficiency (Renal disease > II stage, Child-Plugh score >5)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with minor/moderate/severe stroke
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Circulating/neuroimaging biomarkers and GCS | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by Glasgow Coma Scale (GCS)
Circulating/neuroimaging biomarkers and NIHSS | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by NIHSS scale
Circulating/neuroimaging biomarkers and mRS | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by modified Rankin Scale (mRS)
Circulating/neuroimaging biomarkers and Functional Ambulation Classification | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by Functional Ambulation Classification
Circulating/neuroimaging biomarkers and Ashworth scale | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by Ashworth scale
Circulating/neuroimaging biomarkers and MMSE | 54 months
  Correlation between circulating/neuroimaging biomarkers (GFAP as the only biomarker of brain damage, BDNF and VEGF as markers of neuronal regeneration and plasticity) and functional recovery expressed by MMSE scale

SECONDARY OUTCOMES:
Biomarker curve trend | 54 months
  Estimation of the impact of rehabilitation treatment on the trend of the biomarker curve in patients with ischemic stroke, i.e. how GFAP changes in time after treatment (comparison of GFAP levels between times)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy